CLINICAL TRIAL: NCT03037554
Title: The Effects of Sleepwear With Lateralized Thermal Characteristics on Sleep, Proximal Skin Temperature and Sternal Skin Moisture in Menopausal Women
Brief Title: The Effects of Lateralized Thermal Sleepwear on Sleep, Skin Temperature and Skin Moisture in Menopausal Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical difficulties with ambulatory equipment led to unacceptably high levels of data loss. As we would have had to suspend data collection under Covid precautions in any case, we decided to terminate in March of this year.
Sponsor: St. Peter's Hospital, Albany, NY (Other)
Responsible Party: Principal Investigator, Paul Glovinsky, Ph.D., Clinical Director, St. Peter's Sleep Center, St. Peter's Hospital, Albany, NY
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Lateralized Thermal Sleepwear
Record Dates: First submitted 2017-01-19; First posted 2017-01-31 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Menopause Related Conditions
Keywords: Skin Temperature; Hot Flashes; Sleep Disturbance
MeSH Terms: conditions — Hot Flashes; Parasomnias

STUDY DESIGN:
Intervention Model Description: Hierarchical linear model evaluating repeated measures nested within subjects
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment and sham-control sleepwear will be allocated to subjects in a counterbalanced manner by a study administrator who will not otherwise interact with subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateralized Thermal Sleepwear (Experimental): For two consecutive nights subjects will wear Sleepwear with Lateralized Thermal Characteristics
  Interventions: Device: Sleepwear with Lateralized Thermal Characteristics
- Sham-Lateralized Sleepwear (Sham Comparator): For two consecutive nights subjects will wear Sham-Lateralized Sleepwear
  Interventions: Device: Sham-Lateralized Sleepwear

INTERVENTIONS:
Device: Sleepwear with Lateralized Thermal Characteristics — Subjects will wear sleepwear constructed with insulating fabric on one side and conductive fabric on the other side, arranged bilaterally.
  Arms: Lateralized Thermal Sleepwear
Device: Sham-Lateralized Sleepwear — Subjects will wear sleepwear constructed with two insulating fabrics arranged bilaterally.
  Arms: Sham-Lateralized Sleepwear

SUMMARY:
A home-based, sham-controlled, double-blind, crossover study evaluating the effects of wearing sleepwear with lateralized thermal characteristics on subjective and objective sleep measures, proximal skin temperature, and sternal skin moisture in menopausal women complaining of sleep disturbance and vasomotor symptoms.

DETAILED DESCRIPTION:
Sixteen menopausal women who have given informed consent to participate will be medically screened to rule out physiological sleep disorders. Sleep schedules will be regulated to the average bedtime of a two-week baseline sleep log. Subjects will undergo two two-night, home-based monitoring phases, one an experimental and one a control condition, separated by a washout period of at least five nights. The order of conditions will be counterbalanced between subjects in double-blind fashion. In the experimental condition subjects will wear sleepwear constructed of two fabric types arranged bilaterally, with typical cotton spandex insulating material on one side and specialized conductive material on the other. In the control condition subjects will wear sleepwear that is similarly lateralized in terms of appearance but constructed with typical cotton spandex insulating material on both sides. Ambulatory monitoring will include body position, EEG, actigraphy, skin temperature at multiple proximal sites, and sternal skin moisture. Subjective scales of insomnia severity, menopausal symptoms and sleepwear rating will also be employed.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 months since last menstrual period
* Subjective complaint of sleep disturbance, confirmed by Pittsburgh Sleep Quality Index score greater than 5
* Subjective complaint of at least moderate symptoms of menopause, confirmed by modified Kupperman score greater than 15
* Ability to sleep in the left lateral, right lateral and supine positions

Exclusion Criteria:

* Unable to taper off, with health care provider's agreement, hypnotic or sedative medications, hormone replacement therapy, clonidine, gabapentin, or isoflavones and other botanical compounds used to treat vasomotor symptoms of menopause
* Unable to taper to two or fewer caffeinated beverages per day
* Unable to taper to one or fewer alcoholic beverages per day
* Unable to taper off nicotine in any form
* Unable to taper off recreational drugs
* Subjective sleep, based on two-week sleep logs, averaging less than 4.0 or greater than 7.5 hours per night
* Clinical suspicion of obstructive sleep apnea, periodic leg movements or other significant physiological sleep disturbance
* Known skin allergy to silver, cotton, nylon, surgical tape and other adhesives

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-05-21 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | Two nights in the experimental condition and two nights in the control condition.
  Minutes of sleep of any stage, as scored by conventional criteria, across recording period.
Wakefulness After Sleep Onset | Two nights in the experimental condition and two nights in the control condition.
  Minutes of Wakefulness, as scored by conventional criteria, from first epoch of sleep until end of recording period.
Minutes of non-rapid eye movement (NREM) Stage 1 Sleep | Two nights in the experimental condition and two nights in the control condition.
  Minutes of NREM Stage 1 Sleep, as scored by conventional criteria, across recording period.

SECONDARY OUTCOMES:
Proximal Skin Temperature | Measurements taken every 90 seconds across two-night experimental and control conditions
  Thermochron iButton-derived measurements of skin temperature at bilateral Infraclavicular, Lateral Abdominal and Vastus Lateralis sites

OTHER OUTCOMES:
Position Monitoring | Position sampled every two seconds across two nights in experimental condition and two nights in control condition
  Sleep position recorded by iPhone-based SomnoPose app
Sternal Skin Moisture | Measurements taken every three minutes across two nights in experimental condition and two nights in control condition
  Skin humidity at sternum recorded by specialized Thermochron iButton

CONTACTS AND LOCATIONS:
Overall Officials: Paul Glovinsky, Ph.D., Principal Investigator — St. Peter's Sleep Center
Locations (1):
- St. Peter's Sleep Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No